CLINICAL TRIAL: NCT06717035
Title: Evaluation of Performance of MiYOSMART Photochromic and Clear Spectacle Lenses in Myopic Children.
Acronym: PDIMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Bryan Sim XR, Consultant, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SingaporeNEC
Record Dates: First submitted 2024-11-23; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Myopia; Myopia Progression
Keywords: Myopia; Spectacles; Glasses; Myopia Control; Pediatric; DIMS
MeSH Terms: conditions — Myopia | interventions — Lenses

STUDY DESIGN:
Intervention Model Description: Randomization: 202 children will be recruited at 6 institutions following the rules of inclusion and exclusion criteria. Based on a randomization process defined from the study coordinator, children will be allocated to 2 groups: DIMS and PDIMS. The study will be single blinded, meaning that the investigators are not aware of which type of treatment will be associated with which subjects. Subjects cannot be blinded due to the darkening of PDIMS that allows recognition on the type of lens.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Children on clear DIMS lenses (Active Comparator): 202 children will be recruited at 6 institutions following the rules of inclusion and exclusion criteria. Based on a randomization process defined from the study coordinator, children will be allocated to 2 groups: DIMS and PDIMS. The study will be single blinded, meaning that the investigators are not aware of which type of treatment will be associated with which subjects. Subjects cannot be blinded due to the darkening of PDIMS that allows recognition on the type of lens.
  Interventions: Device: EYE001
- Children on photochromic DIMS lenses (Active Comparator): 202 children will be recruited at 6 institutions following the rules of inclusion and exclusion criteria. Based on a randomization process defined from the study coordinator, children will be allocated to 2 groups: DIMS and PDIMS. The study will be single blinded, meaning that the investigators are not aware of which type of treatment will be associated with which subjects. Subjects cannot be blinded due to the darkening of PDIMS that allows recognition on the type of lens.
  Interventions: Device: EYE001

INTERVENTIONS:
Device: EYE001 — Defocus incorporated multiple segments (DIMS) clear vs DIMS photochromic
  Other Names: Defocus incorporated multiple segments (DIMS) lenses

SUMMARY:
This clinical study aims to evaluate the non-inferiority of the photochromic DIMS spectacles lenses performance (PDIMS) compared to clear DIMS spectacles lenses (DIMS) in myopia management.

DETAILED DESCRIPTION:
Myopia now is recognized as one of the important public health problems and myopia prevention and control has become more important. Various myopia management strategies have been tested in the past for the control of myopia progression in children. In recent years, various optical interventions have also been explored to manage myopia, including the use of optical, pharmaceutical, and lifestyle interventions. Spectacles, atropine eye drops, and outdoor activities have shown some efficacy in slowing myopia progression, but the optimal approach to delaying or preventing the onset of myopia in at-risk populations remains a challenge. These myopia management modalities are often also labelled as invasive and non-invasive methods. One of the non-invasive myopia management modalities includes spectacles.

DIMS spectacle lenses are based on creating myopic defocus at the mid-periphery of the retina which would provide a cue of axial length elongation control. DIMS is a spectacle lens with a central optical zone of 9.4 mm for correcting distance myopic refractive errors and a mid-peripheral 33mm of treatment zone with multiple segments of 1 mm diameter, each segment provides defocus of + 3.5D. 2-year Randomised Controlled Trial (RCT) showed 52% reduction in myopia progression and 62% slow down effect in axial elongation in children wearing DIMS spectacle lenses compared to those on single vision spectacle lens correction at the end of 2-year follow-up in Hong Kong children.

2-years RCT has been conducted using DIMS clear spectacle lenses, however, no studies have been conducted on photochromic and polarized version to show the non-inferiority of sun solutions compared to clear version in myopia management.

This clinical study aims to evaluate the non-inferiority of the photochromic DIMS spectacles lenses performance (PDIMS) compared to clear DIMS spectacles lenses (DIMS) in myopia management.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all the criteria listed to participate in the study:

1. All ethnicities
2. Age between 6 and 15 years
3. Refraction -0.50D till - 7.00D and astigmatism ≤ 3.00D
4. Anisometropia ≤ 3.00D
5. Best corrected monocular distance high contrast VA ≤ 0.10 logMAR
6. Normal Binocular vision (fusion and stereopsis)

Exclusion Criteria

All subjects meeting any of the exclusion criteria at baseline will be excluded from participation:

1. Ocular and systemic abnormalities
2. Children who do not cooperate
3. Binocular vision anomalies (strabismus, suppression)
4. Previous use of myopia management treatment (spectacles, atropine, CLs)
5. Neurological disorders
6. Premature infants
7. Children who do not wear their glasses correctly for intermediate and near vision activities
8. Children who do not meet the inclusion criteria
9. No informed consent given by parents of child for participation in the clinical study
10. Subject is allergic to cycloplegic eye drops

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Comparing photochromic DIMS spectacles lenses performance (PDIMS) versus clear DIMS spectacles lenses (DIMS) | 24 months
  The primary objective of this study is to evaluate the efficacy of photochromic DIMS spectacles lenses performance (PDIMS) compared to clear DIMS spectacles lenses (DIMS) in terms of childhood myopia control (cycloplegic spherical equivalent refraction (SER), axial elongation and choroidal thickness).

SECONDARY OUTCOMES:
Performance of photochromic DIMS spectacles lenses performance (PDIMS) compared to clear DIMS spectacles lenses (DIMS) | 24 months
  To assess the safety, tolerability (quality of life (QoL)), and adaptation to PDIMS lens wear compared to DIMS lens wear.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Change in spherical equivalent and axial length over time for further trials in future
Supporting Information: Study Protocol, CSR
Time Frame: 2025-2026
Access Criteria: Interested investigators
URL: https://www.hoyavision.com/sg/

REFERENCES:
- [Background] Lam CS, Tang WC, Lee PH, Zhang HY, Qi H, Hasegawa K, To CH. Myopia control effect of defocus incorporated multiple segments (DIMS) spectacle lens in Chinese children: results of a 3-year follow-up study. Br J Ophthalmol. 2022 Aug;106(8):1110-1114. doi: 10.1136/bjophthalmol-2020-317664. Epub 2021 Mar 17. PMID 33731364
- [Background] Lam CSY, Tang WC, Tse DY, Lee RPK, Chun RKM, Hasegawa K, Qi H, Hatanaka T, To CH. Defocus Incorporated Multiple Segments (DIMS) spectacle lenses slow myopia progression: a 2-year randomised clinical trial. Br J Ophthalmol. 2020 Mar;104(3):363-368. doi: 10.1136/bjophthalmol-2018-313739. Epub 2019 May 29. PMID 31142465